CLINICAL TRIAL: NCT03550326
Title: Evaluation of Complications During Airway Management: An Observational Prospective Cohort Study
Brief Title: Evaluation of Complications in Airway Management
Acronym: AMC
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principle Investigator, Derince Training and Research Hospital
Other Study IDs: DerinceTRH-05
Record Dates: First submitted 2018-05-27; First posted 2018-06-08 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Airway Complication of Anesthesia; Difficult Intubation
Keywords: anesthesia; difficult airway; supraglottic airway device; difficult intubation; airway complications
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general anesthesia: Patients who undergo general anesthesia and are intubated or inserted airway device will be enrolled. researchers will follow the induction and intubation period and record all the complications due to airway management.
  Interventions: Procedure: airway management

INTERVENTIONS:
Procedure: airway management — patients will be intubated or will be placed an airway device

SUMMARY:
In the current study researchers aim to evaluate the rate of the complication due to airway management (during intubation or placement of supraglottic airway devices)

DETAILED DESCRIPTION:
Airway management is one of the most important subject of anesthesia practice. Airway devices ,helping anesthesiologists to maintain airway safety have many complications. 4 th national audit project (NAP 4) study was designed to evaluate the incidence of the major complication of airway management. Accordingly in current study authors aim to determine the complications and incidence of the complications during airway management.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia
* Patients to whom airway devices will be inserted

Exclusion Criteria:

* Patients who undergo surgery under regional anesthesia
* Patients who undergo surgery under sedation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who undergo surgery under general anesthesia and who intubate/place supraglottic airway device will be recruit for study over a period of six months
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence of the complications due to airway management | 6 months
  researchers will observe the whole patients who undergo general anesthesia and record the data

SECONDARY OUTCOMES:
variety of complications and reasons of the complications | 6 months
  researchers will observe the whole patients who undergo general anesthesia and record the data
preventable reasons of the complications | 6 months
  researchers will observe the whole patients who undergo general anesthesia and record the data
the time at which complications occurs more, during airway management | 6 months
  researchers will observe the whole patients who undergo general anesthesia and record the data

CONTACTS AND LOCATIONS:
Overall Officials: tolga k saracoglu, assoc. prof., Study Director — Sağlık Bilimleri Üniversitesi Kocaeli Derince SUAM
Locations (1):
- Derince Research and Training Hospital, Kocaeli, Turkey (Türkiye)